CLINICAL TRIAL: NCT01430325
Title: Test of Chamber Pressure to Divers and Chamber Attendants: A Blinded Trial to Investigate if "Pressure-familiar" Individuals Can Determine Pressure
Brief Title: Test of Chamber Pressure to Divers and Chamber Attendants
Acronym: TOP-DIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 1023955
Record Dates: First submitted 2011-09-02; First posted 2011-09-08 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2012-12

CONDITIONS: Traumatic Brain Injury
Keywords: Hyperbaric oxygen
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sea Level Equivalent 1.2 atm abs (air) (Sham Comparator): Sham Chamber Session
  Sea Level Equivalent 1.2 atm abs (2.6 psig) breathing regular air 20-chamber excursion
  Interventions: Drug: Sham Chamber Session
- Sea Level Equivalent 1.5 atm abs (O2) (Experimental): Hyperbaric Oxygen (1.5 atm abs)
  Sea Level Equivalent 1.5 atm abs (6.2 psig) breathing 100% oxygen 20-minute chamber excursion
  Interventions: Drug: Hyperbaric Oxygen (1.5 atm abs)
- Altitude Equivalent 1.2 atm abs (air) (Sham Comparator): Sham Chamber Session
  Altitude Equivalent 1.2 atm abs (5.1 psig) breathing regular air 20-minute chamber excursion
  Interventions: Drug: Sham Chamber Session
- Altitude Equivalent 1.5 atm abs (O2) (Experimental): Hyperbaric Oxygen (1.5 atm abs)
  Altitude Equivalent 1.5 atm abs (9.6 psig) breathing 100% oxygen 20-minute chamber excursion
  Interventions: Drug: Hyperbaric Oxygen (1.5 atm abs)

INTERVENTIONS:
Drug: Hyperbaric Oxygen (1.5 atm abs) — Hyperbaric oxygen (100% oxygen) delivered at a chamber pressure of 1.5 atm abs.
  Other Names: HBO2; HBO; HBOT
  Arms: Altitude Equivalent 1.5 atm abs (O2); Sea Level Equivalent 1.5 atm abs (O2)
Drug: Sham Chamber Session — Sham control chamber session: regular air delivered at a chamber pressure of 1.2 atm abs
  Other Names: Sham control; Air pressurization
  Arms: Altitude Equivalent 1.2 atm abs (air); Sea Level Equivalent 1.2 atm abs (air)

SUMMARY:
SCUBA divers and chamber inside attendants will undergo a brief hyperbaric chamber excursion and will be asked to what chamber pressure they were compressed and what gas they breathed.

DETAILED DESCRIPTION:
In clinical trials evaluating hyperbaric oxygen, blinding can be challenging. Options for participant blinding include offering regular air at a lower pressure than the hyperbaric oxygen intervention, or compressing all participants to the same pressure but providing different gas mixes to the active and sham arms.

In some trials of hyperbaric oxygen for brain injury, investigators offer a sham chamber session (regular air at 1.2 atmospheres absolute [atm abs]) compared to the active intervention, hyperbaric oxygen (100% oxygen at 1.5 atm abs). It is unknown whether individuals familiar with pressure changes, such as divers and hyperbaric chamber inside attendants, could discern the difference between these pressures and thereby become unblinded to study allocation.

In this study, 80 experienced divers and chamber inside attendants will be enrolled and randomly assigned to one of four possible chamber pressures and one of two breathing gases. After a brief hyperbaric chamber excursion, they will be asked to what chamber pressure they were compressed and what gas they breathed. If participants can accurately report chamber pressure or breathing gas, pressure-familiar individuals should be excluded from blinded clinical trials of hyperbaric oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Adult, age 18 - 65 years
* Completion of medical history questionnaire without concerns identified for exposure to increased pressure
* Familiarity with atmospheric pressure change:
* Experienced and active hyperbaric chamber inside attendant: more than 50 hyperbaric compressions, with more than 4 have been in the last 4 months; or
* Experienced and active SCUBA diver: more than 20 lifetime compressed gas open water (not swimming pool) dives, with more than 10 in the last 12 months
* Able to equalize middle ear pressure easily

Exclusion Criteria:

* Pregnancy
* Known risk for barotrauma, as identified on the medical history questionnaire, such as:
* Recent (within 12 months) inner ear or sinus surgery
* Spontaneous pneumothorax
* Pulmonary cysts
* Emphysema
* Bullous lung disease
* Chronic obstructive pulmonary disease needing chronic active therapy
* Inability to tolerate chamber confinement or pressure
* Presence of heart failure
* Presence of any implanted electrical device, except hyperbaric-approved pacemakers
* Presence of middle-ear tympanostomy tubes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindell K. Weaver, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (2):
- United States (2):
  - Intermountain Medical Center, Murray, Utah
  - LDS Hospital, Salt Lake City, Utah

REFERENCES:
- [Background] Clarke D. Effective patient blinding during hyperbaric trials. Undersea Hyperb Med. 2009 Jan-Feb;36(1):13-7. PMID 19341123
- [Background] Jansen T, Mortensen CR, Tvede MF. It is possible to perform a double-blind hyperbaric session: a double-blinded randomized trial performed on healthy volunteers. Undersea Hyperb Med. 2009 Sep-Oct;36(5):347-51. PMID 20112525
- [Background] Weaver LK, Hopkins RO, Churchill S, Haberstock D. Double-Blinding is Possible in Hyperbaric Oxygen (HBO2) Randomized Clinical Trials (RCT) Using a Minimal Chamber Pressurization as Control. Undersea Hyperb Med 1997;24(Suppl):36.
- [Result] Weaver LK, Churchill SK, Bell J, Deru K, Snow GL. A blinded trial to investigate whether 'pressure-familiar' individuals can determine chamber pressure. Undersea Hyperb Med. 2012 Jul-Aug;39(4):801-5. PMID 22908836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 82 individuals responded to study announcements and were pre-screened by telephone, of which 25 were deemed ineligible (due to inadequate diving experience). An additional 15 individuals declined to participate (primarily due to scheduling conflicts). 42 divers and chamber inside attendants signed informed consent and participated in the study.
Pre-assignment Details: All participants signing informed consent continued to group assignment.
Groups:
- Altitude Equivalent 1.2 Atm Abs (Air): Altitude Equivalent 1.2 atm abs (5.1 psig) breathing regular air 20-minute chamber excursion
  Sham Chamber Session : Sham control chamber session: regular air delivered at a chamber pressure of 1.2 atm abs
- Altitude Equivalent 1.5 Atm Abs (O2): Altitude Equivalent 1.5 atm abs (9.6 psig) breathing 100% oxygen 20-minute chamber excursion
  Hyperbaric Oxygen (1.5 atm abs) : Hyperbaric oxygen (100% oxygen) delivered at a chamber pressure of 1.5 atm abs.
- Sea Level Equivalent 1.2 Atm Abs (Air): Sea Level Equivalent 1.2 atm abs (2.6 psig) breathing regular air 20-chamber excursion
  Sham Chamber Session : Sham control chamber session: regular air delivered at a chamber pressure of 1.2 atm abs
- Sea Level Equivalent 1.5 Atm Abs (O2): Sea Level Equivalent 1.5 atm abs (6.2 psig) breathing 100% oxygen 20-minute chamber excursion
  Hyperbaric Oxygen (1.5 atm abs) : Hyperbaric oxygen (100% oxygen) delivered at a chamber pressure of 1.5 atm abs.
Period: Overall Study
Arm/Group | Altitude Equivalent 1.2 Atm Abs (Air) | Altitude Equivalent 1.5 Atm Abs (O2) | Sea Level Equivalent 1.2 Atm Abs (Air) | Sea Level Equivalent 1.5 Atm Abs (O2)
Started | 10 | 12 | 8 | 12
Completed | 10 | 12 | 8 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Altitude Equivalent 1.2 Atm Abs (Air) | Altitude Equivalent 1.5 Atm Abs (O2) | Sea Level Equivalent 1.2 Atm Abs (Air) | Sea Level Equivalent 1.5 Atm Abs (O2) | Total
Number analyzed (Participants) | 10 | 12 | 8 | 12 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 8 | 12 | 42
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45 (10) | 49 (7.8) | 47 (9.3) | 45 (13) | 46 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 4 | 10
  Male | 7 | 10 | 7 | 8 | 32
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 8 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Participants Indicating "I do Not Know" on Depth Questionnaire.
Description: Participants indicating "I do not know" on depth questionnaire instead of providing a free response guess.
Time Frame: Within 15 minutes of chamber excursion
Population: All participants who enrolled in the study were analyzed.
Measure: Number; unit: participants
Arm/Group | Altitude Equivalent 1.2 Atm Abs (Air) | Altitude Equivalent 1.5 Atm Abs (O2) | Sea Level Equivalent 1.2 Atm Abs (Air) | Sea Level Equivalent 1.5 Atm Abs (O2)
Number analyzed (Participants) | 10 | 12 | 8 | 12
participants | 7 | 4 | 4 | 4

2. Primary Outcome: Participant Perception of Depth
Description: Mean depth perception for participants providing a free response.
Time Frame: Within 15 minutes of chamber excursion
Population: 23 of 42 participants provided a numerical response. The remainder selected "I do not know."
Measure: Mean (Standard Deviation); unit: fsw
Arm/Group | Altitude Equivalent 1.2 Atm Abs (Air) | Altitude Equivalent 1.5 Atm Abs (O2) | Sea Level Equivalent 1.2 Atm Abs (Air) | Sea Level Equivalent 1.5 Atm Abs (O2)
Number analyzed (Participants) | 4 | 8 | 4 | 7
fsw | 65 (13) | 35 (16) | 23 (12) | 23 (14)

3. Primary Outcome: Participant Perception of Breathing Gas
Description: Percent of participants in each arm guessing that their breathing gas was 100% oxygen.
Time Frame: Within 15 minutes of chamber excursion
Population: 40 of 42 participants provided an answer to this question.
Measure: Number; unit: percentage of participants
Arm/Group | Altitude Equivalent 1.2 Atm Abs (Air) | Altitude Equivalent 1.5 Atm Abs (O2) | Sea Level Equivalent 1.2 Atm Abs (Air) | Sea Level Equivalent 1.5 Atm Abs (O2)
Number analyzed (Participants) | 10 | 11 | 8 | 11
percentage of participants | 80 | 91 | 88 | 67

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time that participants signed consent until they departed after the chamber excursion (approximately 1 hour).
Arm/Group | Altitude Equivalent 1.2 Atm Abs (Air) | Altitude Equivalent 1.5 Atm Abs (O2) | Sea Level Equivalent 1.2 Atm Abs (Air) | Sea Level Equivalent 1.5 Atm Abs (O2)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 1/10 | 0/12 | 0/8 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Altitude Equivalent 1.2 Atm Abs (Air) (N=10) | Altitude Equivalent 1.5 Atm Abs (O2) (N=12) | Sea Level Equivalent 1.2 Atm Abs (Air) (N=8) | Sea Level Equivalent 1.5 Atm Abs (O2) (N=12)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — One participant complained of a slight headache following the chamber excursion, which he attributed to voluntarily skipping meals that day.

LIMITATIONS AND CAVEATS:
Smaller sample size; enrollment was stopped at 42 participants when investigators had exhausted the planned recruitment methods. Very few inside attendants enrolled. Pressures in this study were relatively close.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes